CLINICAL TRIAL: NCT00083993
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Blind Study of Oral CCI-779 Administered in Combination With Letrozole vs. Letrozole Alone as First Line Hormonal Therapy in Postmenopausal Women With Locally Advanced or Metastatic Breast Cancer
Brief Title: Study Evaluating CCI-779 and Letrozole in Post-menopausal Women With Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3066A1-303
Record Dates: First submitted 2004-06-04; First posted 2004-06-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — temsirolimus; WW Domain-Containing Oxidoreductase; Letrozole

INTERVENTIONS:
Drug: Temsirolimus (CCI-779) for 34 months
Drug: Letrozole for 34 months

SUMMARY:
In this clinical research study, postmenopausal subjects with metastatic breast cancer will be given either the combination of temsirolimus (CCI-779) and letrozole or a placebo and letrozole in first-line hormonal treatment. The primary endpoint of this study is to determine overall progression free survival.

Individual subjects will participate in the active treatment phase of the study until disease progression or withdrawal of consent, provided that test article is being tolerated. All subjects will be asked to participate in the long-term follow-up phase of the study, which includes follow-up every 3 months until disease progression (for subjects who withdraw for reasons other than documented progressive disease) or until any new cancer treatment is received, and for survival. The estimated duration of study participation is 34 months.

ELIGIBILITY:
Inclusion Criteria:

* Women aged greater than 18 years.
* Postmenopausal subjects
* Confirmed diagnosis of locally advanced (not amenable to curative surgery and/or radiation) or metastatic breast cancer (Stage 3B or 4 respectively, by American Joint Committee on Cancer Criteria)

Exclusion Criteria:

* Extensive visceral disease
* Subjects with bone as the only site of disease
* Prior radiation therapy to the site of measurable disease for subjects with a solitary measurable lesion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1236
Dates: Start 2004-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To determine overall progression free survival.

SECONDARY OUTCOMES:
To determine safety, survival, health outcomes, prognostic markers and pharmacogenomics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (115):
- United States (101):
  - Hoover, Alabama
  - Huntsville, Alabama
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Burbank, California
  - Campbell, California
  - Fountain Valley, California
  - Gilroy, California
  - Glendora, California
  - Modesto, California
  - Montebello, California
  - Pomona, California
  - Poway, California
  - Sacramento, California
  - San Diego, California
  - Santa Rosa, California
  - Soquel, California
  - Vista, California
  - Lakewood, Colorado
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Lake Worth, Florida
  - Miami Shores, Florida
  - New Port Richey, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Roswell, Georgia
  - Thomasville, Georgia
  - Coeur d'Alene, Idaho
  - Centralia, Illinois
  - Skokie, Illinois
  - Springfield, Illinois
  - Urbana, Illinois
  - Munster, Indiana
  - South Bend, Indiana
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Frederick, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Flint, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Hattiesburg, Mississippi
  - Rolla, Missouri
  - Great Falls, Montana
  - Omaha, Nebraska
  - Carson City, Nevada
  - Lebanon, New Hampshire
  - Belleville, New Jersey
  - Somerset, New Jersey
  - Albuquerque, New Mexico
  - Binghamton, New York
  - East Syracuse, New York
  - New York, New York
  - Nyack, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Gastonia, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Mayfield Heights, Ohio
  - Corvallis, Oregon
  - Portland, Oregon
  - Harrisburg, Pennsylvania
  - Hershey, Pennsylvania
  - Langhorne, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Irving, Texas
  - Tyler, Texas
  - Logan, Utah
  - Ogden, Utah
  - Arlington, Virginia
  - Richmond, Virginia
  - Woodbridge, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
- Canada (14):
  - Calgary, Alberta
  - North Vancouver, British Columbia
  - Richmond, British Columbia
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Hamilton, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Fleurimont, Quebec
  - Lévis, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Wolff AC, Lazar AA, Bondarenko I, Garin AM, Brincat S, Chow L, Sun Y, Neskovic-Konstantinovic Z, Guimaraes RC, Fumoleau P, Chan A, Hachemi S, Strahs A, Cincotta M, Berkenblit A, Krygowski M, Kang LL, Moore L, Hayes DF. Randomized phase III placebo-controlled trial of letrozole plus oral temsirolimus as first-line endocrine therapy in postmenopausal women with locally advanced or metastatic breast cancer. J Clin Oncol. 2013 Jan 10;31(2):195-202. doi: 10.1200/JCO.2011.38.3331. Epub 2012 Dec 10. PMID 23233719